CLINICAL TRIAL: NCT07102719
Title: A Randomized, Open-label, Crossover, Phase 1 Study to Evaluate Pharmacokinetics and Safety of HD-P023 in Comparison With Coadministration of Teneligliptin and Empagliflozin High in Healthy Volunteers
Brief Title: Pharmacokinetics and Safety of HD-P023 and Co-administration of Teneligliptin and Empagliflozin High in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HD-MP-109
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HD-P023 (Experimental): One tablet of HD-P023 by oral
  Interventions: Drug: HD-P023
- Co-administration of Teneligliptin and Empagliflozin High (Active Comparator): One tablet each of Teneligliptin and Empagliflozin High by oral
  Interventions: Drug: Teneligliptin and Empagliflozin

INTERVENTIONS:
Drug: HD-P023 — Single dose administration of HD-P023
  Arms: HD-P023
Drug: Teneligliptin and Empagliflozin — Single does administration of Teneligliptin and Empagliflozin High
  Arms: Co-administration of Teneligliptin and Empagliflozin High

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and safety of HDP023 and coadministration of Teneligliptin and Empagliflozin in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 19 years or older on screening
* Signed informed consent
* Healthy Volunteer
* Other inclusion applies

Exclusion Criteria:

* Clinically relevant/significant findings as evaluated by the investigator
* Other exclusion applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUCt) of Teneligliptin and Empagliflozin | 72 hours
Peak Plasma Concentration (Cmax) of Teneligliptin and Empagliflozin | 72 hours

SECONDARY OUTCOMES:
AUC∞ of Teneligliptin and Empagliflozin | 72 hours
AUCt/AUC∞ of Teneligliptin and Empagliflozi | 72 hours
Tmax of Teneligliptin and Empagliflozin | 72 hours
VZ/F of Teneligliptin and Empagliflozin | 72 hours
CL/F of Teneligliptin and Empagliflozin | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea